CLINICAL TRIAL: NCT06119542
Title: Endothelial Glycocalyx Damage in Major Spine Surgery, as Measured by Circulating Syndecan-1 Levels: a Prospective Observational Pilot Study.(GlycOrtho)
Brief Title: Endothelial Damage in Major Spine Surgery, Measured by Circulating Syndecan-1: an Observational Study.(GlycOrtho)
Acronym: GlycOrtho
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 1064/2021/Oss/IOR
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Spinal Fusion
Keywords: Endothelium; Syndecan-1; Surgery; Glycocalyx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about endothelial damage in major spine surgery, expressed as rise in circulating Syndecan-1.

The main questions it aims to answer are:

* What is the extent of endothelial glycocalyx shedding in major spine surgery?
* Are there differences in different type of surgical populations? (adolescent idiopathic scoliosis, adult degenerative spine disease, oncologic surgery)

To do so, blood samples will be drawn from participants at the following timepoints:

* basal
* after surgery
* if transfusion of Fresh Frozen Plasma: before and after transfusion
* Post-Operative Day 1-2-4

DETAILED DESCRIPTION:
The aim of this study is to gain information about endothelial damage in major spine surgery, expressed as shedding of glycocalyx component Syndecan-1, and subsequent rise of its plasma levels.

This phenomenon has been extensively described in shock states (sepsis, trauma, cardiac arrest ..) but little is known about endothelial damage in elective major surgery.

This study was designed to study the magnitude of Syndecan-1 rise after spine surgery, divided in three main categories: adolescent idiopathic scoliosis, adult degenerative and oncologic surgery.

The investigators were also interested in the effect of Fresh Frozen Plasma transfusion on Syndecan-1 levels, since previous studies have indicated a potential benefit on endothelial integrity.

The results of this study will be used to inform subsequent clinical trials designed to investigate the effect of different intraoperative conducts on endothelial damage.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Major Spine Surgery with estimated blood loss> 25% of total blood volume
* American Society of Anesthesiology status 1-2-3
* Able to comprehend and sign informed consent.
* If age <18 years: parent or legal representative able to comprehend and sign informed consent

Exclusion Criteria:

* Surgery outside of laboratory opening hours
* Patients undergoing spine surgery for genetic syndromes/neuromuscular scoliosis

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will take place in patients undergoing major spine surgery.
  As a secondary analysis, patients will be divided in three major groups:
  * Adolescent idiopathic
  * Adult degenerative spine disease
  * Cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Delta Syndecan-1 before -after surgery | baseline, day 1
  Difference between basal Syndecan-1 level and level at the end of surgery

SECONDARY OUTCOMES:
Post-Operative Syndecan-1 curve | baseline, day 1, day2, day 3, day 5
  Variation of Syndecan-1 levels at post-operative days 1-2-4
Population differences | baseline, day 1, day2, day 3, day 5
  Difference in baseline and post-operative Syndecan-1 levels in different populations

OTHER OUTCOMES:
Thrombomodulin | baseline, day 1, day2, day 3, day 5
  Variations of Thrombomodulin levels
Plasma effect | baseline, day 1
  Difference in Syndecan-1 levels before and after fresh frozen plasma transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Giannone, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Sandra Giannone, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johansson PI, Stensballe J, Ostrowski SR. Shock induced endotheliopathy (SHINE) in acute critical illness - a unifying pathophysiologic mechanism. Crit Care. 2017 Feb 9;21(1):25. doi: 10.1186/s13054-017-1605-5. PMID 28179016
- [Background] Bashandy GM. Implications of recent accumulating knowledge about endothelial glycocalyx on anesthetic management. J Anesth. 2015 Apr;29(2):269-78. doi: 10.1007/s00540-014-1887-6. Epub 2014 Aug 1. PMID 25082728
- [Background] Johansson PI, Haase N, Perner A, Ostrowski SR. Association between sympathoadrenal activation, fibrinolysis, and endothelial damage in septic patients: a prospective study. J Crit Care. 2014 Jun;29(3):327-33. doi: 10.1016/j.jcrc.2013.10.028. Epub 2014 Jan 28. PMID 24581948
- [Background] Milford EM, Reade MC. Resuscitation Fluid Choices to Preserve the Endothelial Glycocalyx. Crit Care. 2019 Mar 9;23(1):77. doi: 10.1186/s13054-019-2369-x. PMID 30850020